CLINICAL TRIAL: NCT02625220
Title: Dispensing Evaluation of Investigational Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-5769
Record Dates: First submitted 2015-11-03; First posted 2015-12-09 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prototype toric lens senofilcon A (Experimental): Subjects will wear the senofilcon A prototype toric contact lens bilaterally for 6-8 days as a daily disposable modality.
  Interventions: Device: Prototype toric lens senofilcon A

INTERVENTIONS:
Device: Prototype toric lens senofilcon A — Investigational prototype

SUMMARY:
Non-randomized, single-masked, 2-visit, bilateral wear, single-arm dispensing study to evaluate the visual acuity, rotational performance, lens fit, stability and subjective characteristics of a senofilcon-based JJVCI investigational toric contact lens design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males or females that are ≥18 years of age and ≤39 years of age.
* The subject must read, understand, and sign the Statement of Informed Consent and receive a fully executed copy of the form.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
* The subject must be a habitual toric contact lens wearer. Habitual wearer is defined as someone who wears toric lenses for at least 6 hours a day, 5 days a week for the past 30 days.
* Subject's vertex corrected spherical component of their distance refraction must be between -1.50 Diopters Sphere (DS) to -4.00 DS (inclusive) in each eye.
* Subject's vertex corrected refractive cylinder must be between -0.75 and -1.50 Diopters Cylinder (DC) (inclusive) in each eye.
* Subject's refractive cylinder axis must be within 180±15° and 90±15° in each eye.
* If needed, the subject must have a wearable pair of spectacles with 20/30 or better vision Ocular Uterque (OU). If spectacles are not needed, the subject must have 20/40 or better vision OU without correction.
* Subject's best corrected distance acuity must be 20/25-2 or better in each eye.

Exclusion Criteria:

* Females who are currently pregnant or lactating.
* Any ocular or systemic allergies or diseases that may contraindicate contact lens wear.
* Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, recurrent herpes simplex/zoster, Sjogren's syndromes, xerophthalmia, acne rosacea, and/or Stevens-Johnson syndromes, by self-report.
* Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g., HIV), by self-report.
* Habitual wearer of extended wear contact lenses.
* Any previous history of ocular and/or refractive surgery (e.g., radial keratotomy, photorefractive keratectomy (PRK), laser-assisted in situ keratomileusis (LASIK), etc.)
* History of seizures.
* Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion by report.
* History of binocular vision abnormality or strabismus, by self-report.
* Habitual wearer of rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
* Employee and family members of employee of investigational clinic (e.g., Investigator, Coordinator, Technician).
* Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
* Any grade 3 or greater slit lamp findings (e.g. edema, corneal neovascularization, corneal staining, tarsal abnormalities, and conjunctival injection) on the FDA classification scale.
* Any history of a contact lens-related corneal inflammatory event within the past year that may contraindicate contact lens wear.
* Any active ocular infection.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Any fluctuations in vision due to clinically significant dry eye or other ocular conditions.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 177 (Actual)
Dates: Start 2015-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Edward S. Wygonik, OD, Jacksonville, Florida
  - The Eye Center, Pembroke Pines, Florida
  - Eye Associates of Winter Park, Winter Park, Florida
  - Eyecare Associates, Bloomington, Illinois
  - Indiana University College of Optometry, Bloomington, Indiana
  - Kannarr Eye Care, Pittsburg, Kansas
  - ABQ Eyecare, Albuquerque, New Mexico
  - Sacco Eye Group, Vestal, New York
  - New Image Eye Center, Springfield, Ohio
  - Professional Vision Care, Westerville, Ohio
  - West Bay Eye Associates, Warwick, Rhode Island
  - Total Eye Care PA, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 177 subjects were enrolled into this study. Of the enrolled subjects, 7 did not meet the eligibility criteria and 170 subjects were dispensed a study lens. Of the dispensed subjects, 7 were discontinued and 163 completed the study.
Groups:
- Prototype Toric Lens Senofilcon A: All subjects in this study were dispensed the prototype toric lens senofilcon A in this study.
Period: Overall Study
Arm/Group | Prototype Toric Lens Senofilcon A
Started | 170
Completed | 163
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 1
Not completed — Study discontinued at site | 2

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed a study lens.
Arm/Group | Prototype Toric Lens Senofilcon A
Number analyzed (Participants) | 170
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.8 (5.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112
  Male | 58
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Native Alaskian | 4
  Asian | 7
  Black or African American | 19
  Native Hawaiian or Other Pacific Islander | 2
  White | 131
  Other | 7
Region of Enrollment [Number; unit: participants]
  United States | 170

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eyes With Monocular Visual Acuity Better Than 20/40
Description: Monocular visual acuity was assessed using distance Snellen visual acuity. Visual Acuity data was dichotomized such that 'response=1' if a subjects has 20/40 or better and 'response=0' if subject has worse than 20/40. The proportion of eyes with 20/40 or better was reported.
Time Frame: 7 day follow-up
Population: The analysis population consists of subjects that completed all study visits without a major protocol deviation (per-protocol). One subject was excluded from the analysis population due to a major protocol deviation.
Measure: Number; unit: proportion of Subject Eyes
Units Other Than Participants: Subject Eyes
Arm/Group | Prototype Toric Lens Senofilcon A
Number analyzed (Participants) | 162
Number analyzed (Subject Eyes) | 324
proportion of Subject Eyes | 1.0

2. Primary Outcome: The Proportion of Eyes With Absolute Rotation Less Than or Equal to 10 Degrees
Description: Absolute rotation was measured using a slit lamp. Absolute rotation measured at 15-minute post insertion was categorized into a binary outcome as 'response=1' if the absolute rotation is less than or equal to 10 degrees or 'response=0' otherwise. The proportion of eyes with absolute rotation less than or equal to 10 degrees was reported.
Time Frame: 15 Minutes Post Insertion
Population: as for outcome 1
Measure: Number; unit: proportion of Subject Eyes
Units Other Than Participants: Subject Eyes
Arm/Group | Prototype Toric Lens Senofilcon A
Number analyzed (Participants) | 162
Number analyzed (Subject Eyes) | 324
proportion of Subject Eyes | 0.993

3. Primary Outcome: Proportion of Subjects Eyes With Lens Stability With Blink Within 5 Degrees
Description: Lens stability with blink was measured using a slit lamp. The rotational stability of the lens during a series of normal (unforced) blinks was measured for both eyes. The data was dichotomized as 'response=1' if the lens stability was less than or equal to 5 degrees or 'response=0' otherwise. The proportion of eyes with rotational stability of 5 degrees or lower was reported.
Time Frame: 15 Minutes Post Insertion
Population: as for outcome 1
Measure: Number; unit: proportion of Subject Eyes
Units Other Than Participants: Subject Eyes
Arm/Group | Prototype Toric Lens Senofilcon A
Number analyzed (Participants) | 162
Number analyzed (Subject Eyes) | 324
proportion of Subject Eyes | 1.0

4. Primary Outcome: Proportion of Subject Eyes With Acceptable Lens Fit
Description: Acceptability of contact lens fit was assessed via slit lamp and was reported as a binary response as Acceptable or Unacceptable. The proportion of eyes with acceptable fit was reported.
Time Frame: 15 Minute Post Insertion
Population: as for outcome 1
Measure: Number; unit: proportion of Subject Eyes
Units Other Than Participants: Subject Eyes
Arm/Group | Prototype Toric Lens Senofilcon A
Number analyzed (Participants) | 162
Number analyzed (Subject Eyes) | 324
proportion of Subject Eyes | 1.0

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study- approximately 2 months
Arm/Group | Prototype Toric Lens Senofilcon A
Serious Adverse Events (participants affected / at risk) | 0/170
Other Adverse Events (participants affected / at risk) | 0/170

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days